CLINICAL TRIAL: NCT05952375
Title: Exploratory Clinical Trial on the Safety, Efficacy, and Pharmacokinetics of XKDCT086 (iPD-1-Claudin18.2-CAR-T) in Claudin 18.2 Positive Advanced Solid Malignant Tumors: a Single Center, Single Arm, Dose-increasing Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XKDCT086
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Gastric Cancer
Keywords: Chimeric Antigen
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- XKDCT086 treatment for patients with Claudin18.2 target positivity (Experimental): Drug: XKDCT086 (chimeric antigen receptor T cell preparation targeting Claudin18.2)
  Dosage form: Cell suspension
  Dose: 30-50mL/bag
  Medication method: intravenous drip
  Frequency: Once
  Interventions: Drug: Chimeric antigen receptor T cell preparation targeting Claudin18.2

INTERVENTIONS:
Drug: Chimeric antigen receptor T cell preparation targeting Claudin18.2 — Chimeric antigen receptor T cell preparation targeting Claudin18.2

SUMMARY:
The goal of this clinical trial is to assessing the safety and tolerability of XKDCT086 cells against recurrent or refractory solid tumors with Claudin18.2 positivity.This experiment proposes to enroll 9-18 patients, the experimental drug is a chimeric antigen receptor T cell preparation targeting Claudin18.2.

DETAILED DESCRIPTION:
This study adopts a single arm, single center, and dose increasing design, using a "3+3" design for dose increasing to evaluate the safety, tolerance, and effectiveness of XKDCT086 cells, as well as to evaluate the pharmacokinetic characteristics of XKDCT086 cells, the correlation between cytokines and efficacy, and immunogenicity.

The experimental process of this study is divided into seven stages: screening period, blood collection period, baseline period, clearance period, study treatment and safety observation period after treatment, follow-up period, and long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age range from 18 to 75 years old (including threshold), regardless of gender;

  2. Patients with advanced solid malignant tumors with positive expression of Claudin 18.2 (including but not limited to gastric cancer, esophageal gastric junction adenocarcinoma, and esophageal adenocarcinoma); And after sufficient treatment, the condition cannot be completely relieved or continue to progress;;

  3. At least one measurable lesion (non lymph node lesion with a length diameter of ≥ 10mm and lymph node lesion with a short diameter of ≥ 15mm) using the RECIST 1.1 standard;

  4. Expected survival time ≥ 12 weeks;

  5. ECOG score 0-1 points;

  6. The laboratory test values conducted for screening must meet the following standards:

Blood routine examination:

WBC ≥ 3.0 × 10^9/L

ANC ≥ 1.5 × 10^9/L

HB ≥ 80g/L (no blood transfusion received within 2 weeks)

PLT ≥ 100 × 10^9/L

Blood biochemical examination:

ALT and AST ≤ 2.5 × ULN (≤ 5 if accompanied by liver metastasis) × ULN

ALB ≥ 30g/L

Serum creatinine ≤ 1.5 × ULN or GFR>50mL/min (GFR=[(140 age) × weight × (0.85 female)]/(72 × Scr)

TBIL ≤ 1.5 × ULN

Coagulation function test:

APTT ≤ 1.5ULN, while INR or PT ≤ 1.5ULN (without receiving anticoagulant therapy)

7. Women of childbearing age must undergo serum pregnancy tests during screening and before receiving clearance treatment, and the results must be negative;

8. If the patient uses the following drugs, the corresponding situation must be met:

Steroids: Treatment doses of steroids must be discontinued 4 weeks before XKDCT086 infusion. However, physiological alternative doses of steroids are allowed: hydrocortisone or equivalent<6-12mg/mm2/day;

Immunosuppression: Any immunosuppressive drug must be stopped at least 4 weeks before enrollment;

9. Voluntarily participate in clinical trials and sign an informed consent form.

Exclusion Criteria:

* 1. Pregnant or lactating women;

  2. Active hepatitis B, hepatitis C or other infectious diseases (syphilis, HIV)

  3. Any active infection that requires antibiotic treatment;

  4. Have received any immune cell therapy within one year;

  5. Those who had received PD-1/PD-L1 Targeted therapy in the past and had serious adverse reactions (the investigator judged whether they were suitable for inclusion);

  6. Have received Targeted therapy drugs of Claudin18.2 in the past;

  7. Inoculate with live vaccines or attenuated live vaccines within 4 weeks before single collection;

  8. Allergic or intolerant to the research drug Tocilizumab, fludarabine, Cyclophosphamide and other anti drenching drugs selected by the researcher;

  9. Uncontrolled cardio cerebral Vascular disease, such as heart failure or others, existed within 6 months before enrollment;

  10. Within the 6 months prior to enrollment in the study, the subjects had a clinically significant history of arrhythmia or were currently in need of treatment β Abnormalities of antiarrhythmic therapy other than receptor blockers or Digoxin and/or conduction drugs, except atrial fibrillation and paroxysmal supraventricular tachycardia;

  11. Left ventricular Ejection fraction (LVEF)<50% at screening;

  12. Patients with active autoimmune diseases, such as systemic lupus erythematosus, within the first 3 months of screening; Those who require continuous medication throughout the entire trial period;

  13. Before single collection, oxygen inhalation is required to maintain a fingertip blood oxygen saturation of ≥ 95%;

  14. Other malignant tumors occurred within 5 years before enrollment, except for cervical Carcinoma in situ, Cutaneous squamous-cell carcinoma or Basal-cell carcinoma which had been treated for radical treatment before;

  15. Suffering from known symptomatic central nervous system (CNS) diseases;

  16. Surgery was performed within 2 weeks prior to single collection and the researchers believe it may affect patient safety;

  17. The maximum target lesion is greater than 40mm;

  18. The widespread metastasis of tumors involving more than two organs may significantly alter the baseline assessment, the researchers believe; Or the tumor progression is rapid, and from enrollment to clearance, the tumor has reached PD;

  19. Those whose hydrothorax and ascites are greater than grade 2 and cannot be controlled by discharge or Diuretic;

  20. Tumor cells infiltrate the central nervous system, and tumor cells are detected in cerebrospinal fluid or detected on cranial imaging;

  21. The subject has unstable or active gastric ulcers or active gastrointestinal bleeding, or other situations that may require emergency treatment during the trial period, including but not limited to gastrointestinal obstruction, perforation, and massive tumor rupture;

  22. The subject has been taking Anticoagulant all the time and cannot stop taking the drug during the whole test process.

  23. Uncontrollable diabetes (Glycated hemoglobin>8%), uncontrolled hypertension (systolic blood pressure/diastolic blood pressure>160mmHg/100mmHg under medication);

  24. Difficult airways (tumor growth obstructs airways or airway deformities, etc.);

  25. People who are allergic to commonly used first aid and Narcotic;

According to the judgment of the researcher, patients who are not suitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AE) | 12 months
  o characterize the safety profile of XKDCT086 in patients with advanced solid tumor

CONTACTS AND LOCATIONS:
Overall Officials: YU cao, MD, Principal Investigator — The Affiliated Hospital of Qingdao University
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China